CLINICAL TRIAL: NCT01267019
Title: Augmenting Social Cognitive Intervention for Veterans With Schizophrenia
Brief Title: Social Cognition Intervention
Acronym: ASCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHBB-004-10S
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Psychosis
Keywords: social cognition; training intervention
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: vivo augmentation (Experimental): social cognitive training with in vivo augmentation
  Interventions: Behavioral: social cognitive training with in vivo augmentation
- Arm 2: social cognitive (Active Comparator): social cognitive training
  Interventions: Behavioral: social cognitive training
- Arm 3: non-social skills (Active Comparator): non-social skills training
  Interventions: Behavioral: non-social skills training

INTERVENTIONS:
Behavioral: social cognitive training with in vivo augmentation — 24 sessions of social cognitive training plus 6 sessions of in vivo exercises
  Arms: Arm 1: vivo augmentation
Behavioral: social cognitive training — 30 sessions of social cognitive training without in vivo exercises
  Arms: Arm 2: social cognitive
Behavioral: non-social skills training — 30 sessions of skills training that has no specific social content
  Arms: Arm 3: non-social skills

SUMMARY:
Veterans with schizophrenia and schizoaffective disorder experience high levels of disability and poor community outcome, and these poor functional outcomes constitute a major public health concern. The treatment of schizophrenia spectrum disorders has shifted fundamentally from a focus on symptom reduction to a focus on recovery and improving aspects of functioning. Needed improvements in community outcome for patients with these disorders will not occur simply through better control of clinical symptoms. Instead, it is necessary to find new treatments that address the key determinants of poor functional outcome, including social cognition. Both basic (non-social) cognition and social cognition are considered key determinants of functional outcome for schizophrenia and schizoaffective disorder. Basic cognition includes the domains of: learning and memory, vigilance / attention, speed of processing, reasoning and problem solving, and working memory. Social cognition generally refers to mental operations that underlie social interactions, including perceiving, interpreting, managing, and generating responses to socially relevant stimuli, including the intentions and behaviors of others. As part of the investigators' previous Merit grant, they have developed a training program for social cognition and are in the process of validating it. Initial results suggest that the program improves performance on measures of social cognition and functional capacity.

In this study, the investigators will evaluate whether adding an in vivo component (training activities that occur in the community) to the current social cognition intervention facilitates generalization of training effects to community outcome and subjective satisfaction. Outcome measures of social cognition and functional capacity will be examined during the 12 week training program, and durability of benefits will be assessed at a 3-month follow up. Generalization to community functioning and subjective satisfaction will be assessed at the end of training and at the 3-month follow up. The investigators will enroll 105 patients across the 5 years of the study with random assignment to training group (social cognition intervention with in vivo exercises, social cognition intervention without in vivo exercises and control). Subjects will receive assessments at baseline, 6 weeks (mid-point), completion of training (12 weeks), and the 3-month follow up.

ELIGIBILITY:
Inclusion Criteria:

All patients must be diagnosed with Schizophrenia, Schizoaffective Disorder, or Psychosis not otherwise specified (NOS) according to Diagnosis and Statistical Manual (DSM-IV) criteria. In addition, the subjects will meet the following criteria:

* Between 18 and 60 years of age
* Estimated premorbid intelligence quota > 70 (based on reading ability)
* Understand spoken English sufficiently to comprehend testing procedures
* Clinically stable (e.g., no inpatient hospitalization in the 8 weeks prior to enrollment, no significant changes in medication in the 4 weeks prior to enrollment, and none anticipated for the 3 months of participation)
* In sufficient health to be able to walk outdoors unaided for at least 15 minutes.

Exclusion Criteria:

* No clinically significant neurological disease as determined by medical history
* No history of serious head injury (e.g., loss of consciousness longer than 1 hour)
* No physical, cognitive, or language impairment of such severity as to adversely affect the validity of data
* No evidence of drug or alcohol dependence in the past six months, and not intoxicated at time of testing based on urine toxicology screen and saliva alcohol test strip. Subjects who test positive will not be disqualified but instead will be asked to return for testing on a different day. However, subjects who test positive on 3 consecutive occasions will be disqualified from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Green, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Derived] Horan WP, Dolinsky M, Lee J, Kern RS, Hellemann G, Sugar CA, Glynn SM, Green MF. Social Cognitive Skills Training for Psychosis With Community-Based Training Exercises: A Randomized Controlled Trial. Schizophr Bull. 2018 Oct 17;44(6):1254-1266. doi: 10.1093/schbul/sbx167. PMID 29300973

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Vivo Augmentation | Arm 2: Social Cognitive | Arm 3: Non-social Skills
Started | 47 | 53 | 53
Completed | 41 | 47 | 47
Not Completed | 6 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Vivo Augmentation | Arm 2: Social Cognitive | Arm 3: Non-social Skills | Total
Number analyzed (Participants) | 41 | 47 | 47 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.3) | 48.8 (9.1) | 46.7 (10.2) | 47.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 21 | 11 | 41
  Male | 32 | 26 | 36 | 94

OUTCOME MEASURES:

1. Primary Outcome: Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT)
Description: A standardized measure of emotion processing. It is scored as a standard score with a population mean of 100 and standard deviation of 15. It can range from 0 to 200. Higher is better.
  Note: Two of the study arms (in vivo and social cognitive training) receive identical procedures and produce identical outcome numbers for the first 6 weeks of the study.
Time Frame: baseline, 6 weeks, 12 weeks, and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Vivo Augmentation | Arm 2: Social Cognitive | Arm 3: Non-social Skills
Number analyzed (Participants) | 41 | 47 | 47
units on a scale
  Baseline | 87.30 (1.12) | 87.30 (1.12) | 88.46 (1.58)
  6 weeks | 89.23 (1.16) | 89.23 (1.16) | 87.61 (1.62)
  12 weeks | 87.84 (1.76) | 89.78 (1.36) | 87.68 (1.62)
  3 months | 86.78 (1.87) | 90.42 (1.46) | 86.51 (1.87)
Statistical Analysis 1: Comparison: Arm 1: Vivo Augmentation vs Arm 2: Social Cognitive vs Arm 3: Non-social Skills; This is a statistical analysis to determine the training effect of social cognitive skills training (in vivo and social cog versus control); Test type: Superiority or Other; p < .05, Mixed Models Analysis

2. Secondary Outcome: The Awareness of Social Inference Test (TASIT)
Description: A measure of mentalizing (i.e., making inferences about other people). It is scored for accuracy in which higher is better. It ranges from 0 - 64.
  Note: Two of the study arms (in vivo and social cognitive training) receive identical procedures and produce identical outcome numbers for the first 6 weeks of the study.
Time Frame: baseline, 6 weeks, 12 weeks, and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Vivo Augmentation | Arm 2: Social Cognitive | Arm 3: Non-social Skills
Number analyzed (Participants) | 41 | 47 | 47
units on a scale
  Baseline | 44.67 (.82) | 44.67 (.82) | 46.79 (.93)
  6 weeks | 45.45 (.77) | 45.45 (.77) | 46.22 (1.04)
  12 weeks | 46.00 (1.24) | 46.91 (1.05) | 46.81 (1.02)
  3 months | 45.83 (1.4) | 46.91 (1.05) | 46.73 (1.00)
Statistical Analysis 1: Comparison: Arm 1: Vivo Augmentation vs Arm 2: Social Cognitive vs Arm 3: Non-social Skills; Test type: Superiority or Other; p < .05, Mixed Models Analysis

3. Secondary Outcome: Profile of Nonverbal Sensitivity (PONS)
Description: A measure of social perception. It is scored as number correct and higher is better. It ranges from 0 - 110.
  Note: Two of the study arms (in vivo and social cognitive training) receive identical procedures and produce identical outcome numbers for the first 6 weeks of the study.
Time Frame: baseline, 6 weeks, 12 weeks, and 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Vivo Augmentation | Arm 2: Social Cognitive | Arm 3: Non-social Skills
Number analyzed (Participants) | 41 | 47 | 47
units on a scale
  baseline | 75.76 (.91) | 75.76 (.91) | 77.41 (1.16)
  6 weeks | 78.90 (.79) | 78.90 (.79) | 79.24 (1.11)
  12 weeks | 76.83 (1.52) | 78.60 (1.04) | 79.89 (1.16)
  3 months | 76.72 (1.94) | 79.28 (1.28) | 80.56 (1.00)
Statistical Analysis 1: Comparison: Arm 1: Vivo Augmentation vs Arm 2: Social Cognitive vs Arm 3: Non-social Skills; Test type: Superiority or Other; p < .05, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Arm 1: Vivo Augmentation | Arm 2: Social Cognitive | Arm 3: Non-social Skills
Serious Adverse Events (participants affected / at risk) | 5/47 | 4/53 | 3/53
Other Adverse Events (participants affected / at risk) | 0/47 | 0/53 | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Vivo Augmentation (N=47) | Arm 2: Social Cognitive (N=53) | Arm 3: Non-social Skills (N=53)
acute exacerbation of symptoms (Psychiatric disorders) | 5 (5) | 3 (3) | 2 (2)
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
diabetic incident (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes